CLINICAL TRIAL: NCT04973111
Title: A Randomized, Double-Blind, Placebo and Comparator-Controlled Crossover Study to Assess Pharmacokinetic and Pharmacodynamic Effects of CT-868 on the Relationship Between Insulin Secretory Response and Ambient Blood Glucose in Obese Male Subjects and Subjects with T2DM
Brief Title: A Study to Assess CT-868 and the Relationship Between Insulin Secretory Response and Ambient Blood Glucose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carmot Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-868-003
Record Dates: First submitted 2021-07-14; First posted 2021-07-22 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Diabetes
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Overweight; Metabolic Diseases; Body Weight
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Overweight; Metabolic Diseases; Body Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CT-868 (Experimental): SC dose of CT-868 Intervention: Drug: CT-868
  Interventions: Drug: CT-868 as SC Injection
- Placebo (Placebo Comparator): SC dose of placebo matching CT-868 dose Intervention: Drug: Placebo
  Interventions: Drug: Placebo as SC Injection
- Active Comparator (Active Comparator): SC dose of Active Comparator Intervention: Drug: Active Comparator
  Interventions: Drug: Active Comparator as SC Injection

INTERVENTIONS:
Drug: CT-868 as SC Injection — CT-868
  Arms: CT-868
Drug: Placebo as SC Injection — Placebo
  Arms: Placebo
Drug: Active Comparator as SC Injection — Active Comparator
  Arms: Active Comparator

SUMMARY:
A Study to Assess the Effect of CT-868 and the Relationship Between Insulin Secretory Response and Ambient Blood Glucose in Obese Male Subjects and Subjects with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Obese Otherwise Healthy Males
* Part 2: Males or Females with T2D
* Part 1: BMI 30.0-35.0, inclusive
* Part 2: BMI 27.0-45.0, inclusive
* 18-65 years old, inclusive
* Stable body weight for 2 months

Exclusion Criteria:

* Significant medical history
* Uncontrolled hypertension
* History of malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Change in insulin secretion rate and ambient glucose levels | Baseline up to 4 days

SECONDARY OUTCOMES:
Change in blood insulin levels at each level of glucose infusion | Baseline up to 4 days
Change in blood glucose levels at each level of glucose infusion | Baseline up to 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Carmot Therapeutics, Inc., a member of the Roche Group
Locations (1):
- Carmot Clinical Research Unit 101, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://carmot-therapeutics.us/